CLINICAL TRIAL: NCT05181345
Title: Effect of Sleep Debt on Neurophysiological Responses to Heat Exposure
Acronym: ChaSPerf
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2021PBMD05; 2021-A02278-33 (Other: IDRCB)
Record Dates: First submitted 2021-12-20; First posted 2022-01-06 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Heat; Excess; Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal sleep first: The night before the first heat exposure, the participants will have a normal night at home.
  The night before the second heat exposure, the participants sleep will be restricted to 3 hours in bed.
  Interventions: Other: Sleep recording (at home); Other: Heat exposure; Other: Normal sleep; Other: Sleep restriction
- Reduced sleep first: The night before the first heat exposure, the participants sleep will be restricted to 3 hours in bed.
  The night before the second heat exposure, the participants will have a normal night at home.
  Interventions: Other: Sleep recording (at home); Other: Heat exposure; Other: Normal sleep; Other: Sleep restriction

INTERVENTIONS:
Other: Sleep recording (at home) — Before both heat exposures, the sleep-wake rhythm will be measured at home for 7 days using actigraphy and a sleep diary that will have been given to him/her during the inclusion visit.
Other: Heat exposure — The subjects will be exposed twice (2 different visits) to heat (45°C; 60-70% humidity rate) for 3 hours in a climate chamber.
  The subjects will be "equipped" with various external sensors allowing the continuous recording of core temperature, mean skin temperature (9 skin measurement points), heart rate, cerebral electrical activity, cerebral oxygenation, skin vascular conductance (blood flow by laser-doppler), blood pressure and skin conductance.
  Neurophysiological and cognitive exploration (NPCE) includes the Stroop test, the Psychomotor Vigilance Task (PVT) and the odd-ball test.
Other: Normal sleep — The night before one of the two heat exposures (first visit for the "Normal sleep first" group and second visit for the "Reduced sleep first" group), the participants will have a normal night at home. The duration and quality of sleep will be measured using a connected headband (Dreem®) allowing for polysomnography.
Other: Sleep restriction — The night before one of the two heat exposures (first visit for the "Reduced sleep first" group and second visit for the "Normal sleep first" group), the participants' sleep will be restricted. The sleep restriction will correspond to a reduced sleep period with a bedtime of 3 hours (04:00 - 07:00). This night of sleep restriction will be carried out in a sleep apartment (at the lab). The duration and quality of sleep will be measured using a connected headband (Dreem®) allowing for polysomnography.

SUMMARY:
Many people are required to work in stressful situations combining sleep debt and hot environmental conditions. If the effect of sleep debt on cognitive performance is proven, this effect could be increased, during heat exposure, through the deleterious effects of sleep debt on thermoregulatory abilities. These alterations may favour the occurrence of accidents.

The changes in cognitive performance induced by hyperthermia are also poorly characterised and often not dissociated from the effects of dehydration. Little is known about the effects of the combination of sleep debt and heat exposure on mental performance. Describing and understanding the alterations induced by this combined situation could provide a better understanding of the mechanisms explaining the deterioration of performance in hot conditions and promote the development of appropriate countermeasures.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 35 years old
* Body Mass Index between 18 and 27 kg/m2
* Body weight ≥ 54 kg

Exclusion Criteria:

* Presence or history of medical pathology (cardiological, renal, hepatic, cutaneous, intestinal, neurological...)
* Presence of a significant deviation from the normal values observed on the electrocardiogram
* History of heat stroke
* Known intolerance to heat (e.g. migraine sufferers)
* Presence of a contraindication to blood sampling, notably low venous capital, belonephobia
* Inability to ingest a capsule or refusal of the rectal probe
* Habitual consumption of caffeine > 500 mg per day
* Alcohol consumption greater than the equivalent of 3 glasses of wine per week
* Consumption of narcotics
* Smoking > 0.5 packet of cigarettes per day
* Undergoing habitual medication
* Pregnant or breastfeeding woman

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will be composed of healthy young male and female.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Number of errors at the Stroop test | Through study completion (25 months)
  Written color names that differ from the color ink they are printed on will be displayed on a computer screen. In the first trial, the participant must say the written word. In the second trial, the participant must name the ink color instead. The higher the number of correct answers, the higher the score.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recherche Biomédicale des Armées, Brétigny-sur-Orge, France

IPD SHARING:
Plan to Share IPD: Undecided